CLINICAL TRIAL: NCT06703086
Title: Gene Modulation of NLRP3, IL-1β and TNF-α in Peripheral Blood of Patients With Exogenous Obesity Treated With Berberine
Acronym: Obesity-Berber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Modesto Gómez López, Ph.D., Molecular Biologist,, National Polytechnic Institute, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.ESM.CE-01/7-12-2015
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Overweight; Berberine
Keywords: Obesity; Overweight; Berberine
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Phase three clinical trial with three intervention groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nutritional plan only (Active Comparator): Nutritional plan according to your caloric requirements for lifestyle
  Interventions: Behavioral: nutritional plan
- Nutritional plan and moderate aerobic exercise (Active Comparator): nutritional plan and controlled moderate aerobic exercise that will consist of a goal of 10,000 steps or 150 minutes per week
  Interventions: Behavioral: nutritional plan; Behavioral: controlled moderate aerobic exercise
- Berberine, nutritional plan and moderate exercise (Experimental): nutritional plan, moderate aerobic exercise and the phytopharmaceutical Berberine 500 mg every 8 hours for 3 months.
  Interventions: Dietary Supplement: Berberine Hydrochloride group; Behavioral: nutritional plan; Behavioral: controlled moderate aerobic exercise
- No intervention (No Intervention): patients who met the inclusion criteria but did not receive treatment or intervention, only somatometry and blood samples were taken.

INTERVENTIONS:
Dietary Supplement: Berberine Hydrochloride group — The patient will be given a nutritional plan, moderate aerobic exercise with a goal of 10,000 steps or 150 min per week; and the phytopharmaceutical Berberine will be taken 3 tablets ( 500 mg) every 8 hours for 3 months.
  Arms: Berberine, nutritional plan and moderate exercise
Behavioral: nutritional plan — nutritional plan according to your caloric requirements for lifestyle change and you will be scheduled biweekly for 3 months
  Arms: Berberine, nutritional plan and moderate exercise; Nutritional plan and moderate aerobic exercise; Nutritional plan only
Behavioral: controlled moderate aerobic exercise — controlled moderate aerobic exercise that will consist of a goal of 10,000 steps or 150 minutes per week.
  Arms: Berberine, nutritional plan and moderate exercise; Nutritional plan and moderate aerobic exercise

SUMMARY:
The patients will be invited to participate in a research study aimed at determining the Gene Modulation of NLRP3, IL-1β and TNFα in peripheral blood of patients with exogenous obesity treated with berberine.

DETAILED DESCRIPTION:
The study will take 6 months in total, in this study will participate patients with exogenous obesity, which is defined as an abnormal accumulation of fat that can be detrimental to health. After the evaluation it will be determined if you meet the section criteria to be able to participate in the study. The patients will be randomly assigned to a group which may be:

Group I. The investigator will give a nutritional plan according to your caloric requirements for lifestyle change and the patients will be scheduled biweekly for 3 months to assess your weight, height, body mass index and percentages of fat or muscle.

Group 2. The investigator will be given a nutritional plan and controlled moderate aerobic exercise that will consist of a goal of 10,000 steps or 150 minutes per week.

The patient will be given a lifestyle change plan in accordance with their nutritional requirements.

Group 3. The investigator will give a nutritional plan, moderate aerobic exercise with a goal of 10,000 steps or 150 min per week; and the phytopharmaceutical Berberine will take 3 tablets every 8 hours for 3 months.

Biweekly sessions will be carried out for 3 months, then monthly for 6 months; blood samples will be taken at the beginning of the study, that is, after the informed consent, at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with BMI ≥ 30kg/m2

  * With risk factors for type 2 diabetes (history of diabetic parents or siblings, sedentary habits)
  * Fasting blood glucose ≤ 126 mg/dL or glycosylated hemoglobin < 6.5%
  * Controlled arterial hypertension
  * >18 years of age
  * Accept and sign the informed consent

Exclusion Criteria:

* • Pregnancy patients

  * Diabetics patients
  * Presenting any serious adverse effect
  * Patients who decide to withdraw from the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
To determine the effects of Berberine on the gene modulation of NLRP3, in peripheral blood of patients with exogenous obesity | From enrollment to the end of treatment at 3 months
  Extraction of total RNA by TRIzol®Reagent and Real-time polymerase chain reaction, qRT-PCR
To determine the effects of Berberine on the gene modulation of IL-1β in peripheral blood of patients with exogenous obesity | "From enrollment to the end of treatment at 3 months
  Extraction of total RNA by TRIzol®Reagent and Real-time polymerase chain reaction, qRT-PCR
To determine the effects of Berberine on the gene modulation of TNFα in peripheral blood of patients with exogenous obesity | From enrollment to the end of treatment at 3 months
  Extraction of total RNA by TRIzol®Reagent and Real-time polymerase chain reaction, qRT-PCR in peripheral blood

SECONDARY OUTCOMES:
Weight | the first 3 months every 2 weeks, then every month thereafter until 6 months are completed
  The weight will be taken on a scale calibrated in kilograms.
Body mass index | Body mass index will be taken every two weeks for 3 months and then every month for 3 months to complete 6 months.
  The body mass index was calculated by dividing the weight in kilograms by the square of the height in meters.
Percentage of body fat | It will be taken every two weeks for 3 months and then every month for 3 months to complete 6 months.
  Instrument: Body composition analyzer (InBody770).
  • The measurement was expressed in Kg, with a precision of 0.1 kg. It was determined with the body analyzer, programmed with the required parameters (age, sex, height, among others).
Percentage of visceral fat | To be taken every two weeks for the first 3 months and then every month for three months to complete 6 months of follow-up.
  * Instrument: Body composition analyzer (InBody770).
  * The measurement was expressed in Kg, with a precision of 0.1 kg. It was determined with the body analyzer, programmed with the required parameters (age, sex, height, among others).
Height | Height will be measured every two weeks for 3 months and then every month for 3 months to complete the 6 months follow-up.
  It was defined as the distance between the vertex and the support plane.
  * Instrument: Stadiometer (Seca mod. 208).
  * The measurement was expressed in cm with a precision of 1 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia-Mabel PV PhD Nadia Mabel Pérez Vielma, PhD, Study Director — 044-5520583053

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chuang TY, Wu HL, Min J, Diamond M, Azziz R, Chen YH. Berberine regulates the protein expression of multiple tumorigenesis-related genes in hepatocellular carcinoma cell lines. Cancer Cell Int. 2017 May 30;17:59. doi: 10.1186/s12935-017-0429-3. eCollection 2017. PMID 28572744
- [Result] Wei W, Zhao H, Wang A, Sui M, Liang K, Deng H, Ma Y, Zhang Y, Zhang H, Guan Y. A clinical study on the short-term effect of berberine in comparison to metformin on the metabolic characteristics of women with polycystic ovary syndrome. Eur J Endocrinol. 2012 Jan;166(1):99-105. doi: 10.1530/EJE-11-0616. Epub 2011 Oct 21. PMID 22019891
- [Result] Ali AT, Hochfeld WE, Myburgh R, Pepper MS. Adipocyte and adipogenesis. Eur J Cell Biol. 2013 Jun-Jul;92(6-7):229-36. doi: 10.1016/j.ejcb.2013.06.001. Epub 2013 Jun 14. PMID 23876739
- [Result] Sarjeant K, Stephens JM. Adipogenesis. Cold Spring Harb Perspect Biol. 2012 Sep 1;4(9):a008417. doi: 10.1101/cshperspect.a008417. PMID 22952395
- [Result] Merino M, Briones L, Palma V, Herlitz K, Escudero C. Role of adenosine receptors in the adipocyte-macrophage interaction during obesity. Endocrinol Diabetes Nutr. 2017 Jun-Jul;64(6):317-327. doi: 10.1016/j.endinu.2017.03.010. Epub 2017 May 16. English, Spanish. PMID 28604342
- [Result] Fruh SM. Obesity: Risk factors, complications, and strategies for sustainable long-term weight management. J Am Assoc Nurse Pract. 2017 Oct;29(S1):S3-S14. doi: 10.1002/2327-6924.12510. PMID 29024553
- [Result] Siani A, Cappuccio FP, Barba G, Trevisan M, Farinaro E, Lacone R, Russo O, Russo P, Mancini M, Strazzullo P. The relationship of waist circumference to blood pressure: the Olivetti Heart Study. Am J Hypertens. 2002 Sep;15(9):780-6. doi: 10.1016/s0895-7061(02)02976-x. PMID 12219872
- [Result] Peralta-Romero Jde J, Gomez-Zamudio JH, Estrada-Velasco B, Karam-Araujo R, Cruz-Lopez M. [Genetics of pediatric obesity]. Rev Med Inst Mex Seguro Soc. 2014;52 Suppl 1:S78-87. Spanish. PMID 24866313
- [Result] Al-Goblan AS, Al-Alfi MA, Khan MZ. Mechanism linking diabetes mellitus and obesity. Diabetes Metab Syndr Obes. 2014 Dec 4;7:587-91. doi: 10.2147/DMSO.S67400. eCollection 2014. PMID 25506234
- [Result] Heilbronn LK, Campbell LV. Adipose tissue macrophages, low grade inflammation and insulin resistance in human obesity. Curr Pharm Des. 2008;14(12):1225-30. doi: 10.2174/138161208784246153. PMID 18473870

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-08-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT06703086/Prot_SAP_000.pdf
  • Informed Consent Form (2015-08-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT06703086/ICF_001.pdf